CLINICAL TRIAL: NCT02015208
Title: A Phase I/II Trial of Ruxolitinib (Jakafi) in Patients With Chronic Lymphocytic Leukemia Who Are Unfit for Conventional First-line Therapy Due to Age or 17p Deletions
Brief Title: Ruxolitinib in the Treatment of Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINC424XCA03T
Record Dates: First submitted 2013-12-03; First posted 2013-12-19 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL; cytokine signaling; signal transduction inhibitors; elderly; p53
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ruxolitinib (Experimental): Ruxolitinib will be administered over a 28-day cycle, which will be repeated 6 more times in the absence of intolerable toxicity, disease progression, patient withdrawal of consent, or investigator decision to end therapy. The dose and schedule have been adapted from the product monograph for myelofibrosis. The starting dose will be 20 mg orally twice a day with normal .platelet and absolute neutrophil counts and no hepatic and renal impairment.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — 20 mg orally on day 1 to 21 of each 28 day cycle. Number of Cycles: 7 or until progression or unacceptable toxicity develops.
  Other Names: jakafi

SUMMARY:
The purpose of this study is to determine if Ruxolitinib, an inhibitor of cytokine-signaling, is effective in the treatment of patients with Chronic Lymphocytic Leukemia for whom conventional chemotherapy is either too toxic or ineffective.

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia (CLL) is the commonest leukemia in adults and, until recently, had limited treatment options. However, the combination of fludarabine, cyclophosphamide, and rituximab (FCR) produces impressive clinical responses and prolongs survival of many CLL patients with symptomatic disease. Unfortunately, FCR is a toxic regimen that cannot generally be tolerated by patients over the age of 65 years who constitute more than 70% of the CLL patient population. In addition, FCR is contraindicated in patients whose leukemia cells harbor deletions of chromosome 17, where the tumor suppressor p53 is located, because such cells are intrinsically resistant to genotoxic drugs. This group constitutes 10-15% of patients of all ages who require first-line therapy. Better therapies for these two large groups of patients are needed.

The initiating event in CLL is thought to be genetic damage to a class of B lymphocytes that prevents proper functioning of apoptotic pathways. However, disease progression is driven by signals from the proliferation centers in tumor microenvironments where circulating CLL cells originate. Signals that cause CLL cells to proliferate include antigens that activate B-cell receptors (BCRs), Toll-like receptor ligands, chemokines, and cytokines. CLL cells that respond strongly to these microenvironmental signals exhibit more aggressive clinical behavior and resistance to cytotoxic drugs. These observations have motivated the use of signal transduction inhibitors to treat CLL and initial results of targeting kinases in the BCR-signaling cascade, such as Bruton's Tyrosine Kinase (BTK), suggest this strategy is effective and likely to change the treatment paradigm for CLL.

BCR signaling is not the only driver of CLL proliferation in vivo. Cytokines and chemokines in the tumor microenvironment activate Janus Kinases (JAKs) and mediate many of the pathological features of CLL cells. Cytokine signaling pathways have been shown to be rewired in aggressive tumor cells to support rapid growth and will eventually overcome the effects of inhibiting BCR-signaling. Preclinical findings suggest that JAK inhibitors will also have a place in the treatment of CLL.

Based on this strong theoretical rationale and pre-clinical evidence, along with its known toxicity profile, Ruxolitinib is expected to have significant activity with limited toxicity as a single agent in CLL. This trial is designed to investigate the efficacy and toxicity of Ruxolitinib in patients who are otherwise unfit for first-line therapy with FCR.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 65 years unless a 17p deletion is present in more than 20% of circulating tumor cells, in which case age can be younger than 65 years.
2. Diagnosis of CLL meeting published diagnostic criteria.
3. CLL requiring treatment on the basis of National Cancer Institute (NCI) working group criteria.
4. Not previously treated with cytotoxic drugs or antibodies but may have received glucocorticoid monotherapy, local radiation, or splenectomy.
5. Unfit for full dose FCR chemotherapy.
6. Platelets >50x10**9/L. Neutrophils>.75x10**9/L.
7. At least 1 lymph node >1.5 cm or splenomegaly as detected by CT scan.

Exclusion Criteria:

1. Fit for full-dose FCR as initial treatment.
2. Progressive multifocal leukoencephalopathy (PML).
3. Clinically significant bacterial, fungal, parasitic or viral infection, which require therapy.
4. Richter's transformation or prolymphocytic leukemia.
5. Uncontrolled autoimmune hemolytic anemia or idiopathic thrombocytopenia purpura.
6. Prior exposure to chemotherapy for CLL with the exception of glucocorticoids, local radiation, or splenectomy.
7. History of prior malignancy, with the exception of the following: i. Malignancy treated with curative intent and with no evidence of active disease for more than 2 years. ii. Adequately treated skin cancer. iii. Adequately treated cervical carcinoma in situ.
8. Currently active clinically significant cardiovascular disease.
9. History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
10. Renal failure requiring dialysis and patients with moderate and severe renal impairment with platelet counts less than 100,000/ml.
11. Hepatic impairment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Clinical response rate | at 7 months

SECONDARY OUTCOMES:
number of patients with adverse events | participants will be followed for an average of 8 months

OTHER OUTCOMES:
Effects of ruxolitinib on immune and leukemia cell numbers, JAK signaling, and circulating cytokine levels | within 6 months of completing enrollment

CONTACTS AND LOCATIONS:
Overall Officials: David E Spaner, MD, PhD, Principal Investigator — Sunnybrook Health Sciences Center
Locations (1):
- Sunnybrook Odette Cancer Center, Toronto, Ontario, Canada

REFERENCES:
- [Background] Tomic J, Lichty B, Spaner DE. Aberrant interferon-signaling is associated with aggressive chronic lymphocytic leukemia. Blood. 2011 Mar 3;117(9):2668-80. doi: 10.1182/blood-2010-05-285999. Epub 2011 Jan 4. PMID 21205928
- [Derived] Xia M, Luo TY, Shi Y, Wang G, Tsui H, Harari D, Spaner DE. Effect of Ibrutinib on the IFN Response of Chronic Lymphocytic Leukemia Cells. J Immunol. 2020 Nov 15;205(10):2629-2639. doi: 10.4049/jimmunol.2000478. Epub 2020 Oct 16. PMID 33067379